CLINICAL TRIAL: NCT03836131
Title: Rate of Cancer of Granular Mixed Laterally Spreading Tumors (GM-LST): A Restrospective Multicentric Analysis
Brief Title: Rate of Cancer of Granular Mixed Laterally Spreading Tumors (GM-LST)
Acronym: LST GM
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 767
Record Dates: First submitted 2019-02-08; First posted 2019-02-11 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Colorectal cancer (CRC) is the third most common cancer in men and the second in women worldwide, with 1.65 million new cases and almost 835,000 deaths in 2015. CRC is still a major cause of mortality associated with cancer, although the wide spread of the screening program has led to a reduction in the mortality rate compared to the last decades.

CRCs derive from precancerous lesions that may be polypoid or non-polypoid according to the Paris classification. Thus, resection in an early stage could led to a CRC mortality reduction.

Laterally spreading tumors (LST) are non-polypoid lesions of at least 1 cm in diameter that have lateral growth rather than upward or downward growth.

The prevalence of LSTs ranges from 1 to 6% of all colorectal lesions. LSTs can be divided into two groups: granular LSTs, which include homogeneous and granular mixed forms and non-granular (NG) LSTs, which include pseudo-depressed and flat-elevated forms.

Histologically, 90% of LSTs are adenomas and having a low incidence of invasive neoplasia, these lesions can be removed endoscopically.

However, as evidenced by a recent meta-analysis published by Bogie Roel MM et al on Endoscopy, the type of LST and the distal or proximal colonic localization could represent predictors of submucosal invasion and could simplify the therapeutic decision for the removal of these lesions. GM-LSTs and pseudo-depressed NG-LSTs predominantly localize in the distal portion of the colon and have a submucosal invasion rate of 10,5% and 31,6% respectively.

LSTs can be removed both through endoscopic mucosal resection (EMR) and endoscopic submucosal dissection (ESD). The main limitation of EMR is that large lesions require a piecemeal approach, resulting in a non-optimal histological evaluation and a high risk of recurrence. ESD instead allows a higher rate of en bloc resections, thus resulting more curative and reducing the risk of having partial and incomplete resections, which can lead to disease recurrence/non curative resection.

LST-GM are characterized by the presence of a granular appearance with a main nodule and represent approximately 1/4 of the LSTs. There are no guidelines indicating the proper resective technique of these lesions.

The European Society of Gastrointestinal Endoscopy (ESGE) suggests to consider ESD for the removal of colorectal lesions that are > 20 mm in size, with a depressed and irregular morphology or a non-granular surface pattern, as these lesions have a high probability of having a limited submucosal invasion. Moreover ESD can be used to treat lesions that cannot be completely removed with standard polypectomy or EMR.

The investigators propose to perform a multicenter retrospective observational study to define the percentage of cancer in patients with GM-LSTs treated with endoscopic resection in order to evaluate the correlation between pre-resection and post-resection characteristics, defining the best therapeutic approach (en bloc or piecemeal) and avoiding incomplete endoscopic resections or unnecessary surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* LST-GM defined according to Paris classification
* Agree to receive follow up phone calls

Exclusion Criteria:

* Evidence of familial adenomatous polyposis or inflammatory bowel diseases
* Deep submucosal invasion diagnosed by distorted pit pattern (Kudo's type V)
* Poor general clinical condition (American Society of Anesthesiologists score ≥3)
* Coagulation disorders
* Pregnancy and breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a multicenter retrospective observational study. All consecutive patients with GM-LST, who underwent endoscopic resection from, will be enrolled in the study.
  For each procedure LST size, nodule size, location, type of technique used for removal (EMR, ESD, hybrid ESD), type of removal (piecemeal or en bloc), histological examination, possible surgical intervention (and attached histological examination of the operative piece) and possible relapses will be reported.
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2018-12-31 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
The percentage of cancer in patients with GM-LSTs treated with endoscopic resection. | 12 Months

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Humanitas Research Hospital, Milan
  - Humanitas Research Hospital, Rozzano

REFERENCES:
- [Derived] D'Amico F, Amato A, Iannone A, Trovato C, Romana C, Angeletti S, Maselli R, Radaelli F, Fiori G, Viale E, Di Giulio E, Soriani P, Manno M, Rondonotti E, Galtieri PA, Anderloni A, Fugazza A, Ferrara EC, Carrara S, Di Leo M, Pellegatta G, Spadaccini M, Lamonaca L, Craviotto V, Belletrutti PJ, Hassan C, Repici A; Bowell Group. Risk of Covert Submucosal Cancer in Patients With Granular Mixed Laterally Spreading Tumors. Clin Gastroenterol Hepatol. 2021 Jul;19(7):1395-1401. doi: 10.1016/j.cgh.2020.07.024. Epub 2020 Jul 17. PMID 32687977